CLINICAL TRIAL: NCT03188822
Title: A Prospective, Randomized, Controlled Trial of Steroid Delivery to the Frontal Sinus Opening With a Bioabsorbable Steroid Releasing Implant vs. a Bioabsorbable Nasal Dressing With Added Steroid
Brief Title: Steroid Delivery to the Frontal Sinus Opening With a Bioabsorbable Implant vs. a Bioabsorbable Nasal Dressing
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study enrollment was too slow to complete the study in a reasonable time
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Li-Xing Man, Assistant Professor, University of Rochester
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RSRB 00058385
Record Dates: First submitted 2017-06-13; First posted 2017-06-15 (Actual); Results first posted 2021-12-03 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2022-12

CONDITIONS: Chronic Rhinosinusitis (Diagnosis)
MeSH Terms: conditions — Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Bioabsorbable steroid releasing sinus implant & nasal dressing impregnated with steroid (Experimental): Patients will undergo bilateral endoscopic sinus surgery which will include bilateral frontal sinusotomy of Draf 2a or 2b type as previously described in the literature. At the conclusion of the procedure, if the patient still meets all inclusion criteria, one frontal sinus will be randomly assigned using the envelop method to receive a bioabsorbable steroid releasing implant and the other frontal sinus will receive a bioabsorbable nasal dressing impregnated with steroid
  Interventions: Device: Bioabsorbable steroid releasing sinus implant; Device: Bioabsorbable nasal dressing impregnated with steroid

INTERVENTIONS:
Device: Bioabsorbable steroid releasing sinus implant — After completion of indicated frontal sinus surgery, patients will have a bioabsorbable steroid releasing implant placed in the frontal sinus opening, which will remain in place for 14 days.
Device: Bioabsorbable nasal dressing impregnated with steroid — After completion of indicated frontal sinus surgery, patients will have a bioabsorbable nasal dressing impregnated with steroid placed in the frontal sinus opening, which will remain in place for 14 days.

SUMMARY:
The purpose of this study is to compare how two different post-surgical treatments that both deliver steroids to the frontal sinus opening affect your healing after frontal sinus surgery.

DETAILED DESCRIPTION:
This is a single center, randomized & controlled trial comparing the efficacy of the Propel mini stent or Propel contour stent vs. Nasopore impregnated with Triamcinolone Acetonide at reducing frontal sinus opening stenosis and polypoid edema after endoscopic sinus surgery in patients with chronic rhinosinusitis with polyposis. Eligible subjects who undergo standard of care bilateral frontal sinusotomy will have each frontal sinus randomly assigned to either a Propel mini or contour steroid eluding stent or a Nasopore nasal dressing impregnated with 2.5 ml of Triamcinolone Acetonide 40 mg/ml. Specific Propel stent will be chosen based on the shape of frontal sinus opening and best fit as decided by the operating Surgeon. Patients will be reassessed on approximately post-operative day 7, 14, 30, 90 days, 6 months, and 12 months at their standard of care follow-up visits. On the day 14 visit, the frontal sinus Propel stent and Nasopore will be completely removed per Standard of care. Video will be taken of the frontal sinus opening, and assessed for scarring/adhesions, presence of polypoid edema, frontal sinus patency, need for oral steroids or other interventions. Additionally, endoscopic scoring of frontal sinus by the above measures will be evaluated by 2 independent sinus surgeon reviewers. The reviewers will also be asked to rank the two frontal sinus openings as better, same or worse, compared to the opposite side

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 and older
* Diagnosis of chronic rhinosinusitis with nasal polyps based on the American Academy of Otolaryngology-Head and Neck Surgery guidelines
* Patient scheduled for bilateral endoscopic sinus surgery with evidence of bilateral frontal sinus disease based on Computed Tomography (Lund-Mackay score greater than or equal to 1)
* At the time of surgery bilateral frontal sinusotomy of type Draf 2a or 2b was performed using the same technique on both sides
* Bilateral endoscopic sinus surgery performed successfully without complication
* Frontal sinus opening diameter greater than 4.0 mm achieved (4 mm olive tipped suction easily passed into frontal sinus)

Exclusion Criteria:

* Any patient who had frontal sinus surgery for tumor
* Allergy to mometesone and/or triamcinolone
* Frontal sinusotomy type Draf 1 or Draf 3 performed
* One or both frontal sinus openings not amenable to implant placement
* Patients with chronic oral steroid dependent conditions
* Invasive fungal sinusitis
* Immune deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-08-25 (Actual); Primary Completion 2021-09-28 (Actual); Study Completion 2021-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Li-Xing Man, MSc, MD, MPA, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Department of Otolaryngology Head and Neck Surgery, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosenfeld RM, Piccirillo JF, Chandrasekhar SS, Brook I, Ashok Kumar K, Kramper M, Orlandi RR, Palmer JN, Patel ZM, Peters A, Walsh SA, Corrigan MD. Clinical practice guideline (update): adult sinusitis. Otolaryngol Head Neck Surg. 2015 Apr;152(2 Suppl):S1-S39. doi: 10.1177/0194599815572097. PMID 25832968
- [Background] Fokkens WJ, Lund VJ, Mullol J, Bachert C, Alobid I, Baroody F, Cohen N, Cervin A, Douglas R, Gevaert P, Georgalas C, Goossens H, Harvey R, Hellings P, Hopkins C, Jones N, Joos G, Kalogjera L, Kern B, Kowalski M, Price D, Riechelmann H, Schlosser R, Senior B, Thomas M, Toskala E, Voegels R, Wang de Y, Wormald PJ. EPOS 2012: European position paper on rhinosinusitis and nasal polyps 2012. A summary for otorhinolaryngologists. Rhinology. 2012 Mar;50(1):1-12. doi: 10.4193/Rhino12.000. PMID 22469599
- [Background] Ragab SM, Lund VJ, Scadding G, Saleh HA, Khalifa MA. Impact of chronic rhinosinusitis therapy on quality of life: a prospective randomized controlled trial. Rhinology. 2010 Sep 1;48(3):305-11. doi: 10.4193/Rhin08.137. PMID 21038021
- [Background] Chandra RK, Palmer JN, Tangsujarittham T, Kennedy DW. Factors associated with failure of frontal sinusotomy in the early follow-up period. Otolaryngol Head Neck Surg. 2004 Oct;131(4):514-8. doi: 10.1016/j.otohns.2004.03.022. PMID 15467628
- [Background] Valdes CJ, Bogado M, Samaha M. Causes of failure in endoscopic frontal sinus surgery in chronic rhinosinusitis patients. Int Forum Allergy Rhinol. 2014 Jun;4(6):502-6. doi: 10.1002/alr.21307. Epub 2014 Mar 10. PMID 24616299
- [Background] DeConde AS, Smith TL. Outcomes After Frontal Sinus Surgery: An Evidence-Based Review. Otolaryngol Clin North Am. 2016 Aug;49(4):1019-33. doi: 10.1016/j.otc.2016.03.024. PMID 27450618
- [Background] Rowe-Jones JM, Medcalf M, Durham SR, Richards DH, Mackay IS. Functional endoscopic sinus surgery: 5 year follow up and results of a prospective, randomised, stratified, double-blind, placebo controlled study of postoperative fluticasone propionate aqueous nasal spray. Rhinology. 2005 Mar;43(1):2-10. PMID 15844495
- [Background] Wright ED, Agrawal S. Impact of perioperative systemic steroids on surgical outcomes in patients with chronic rhinosinusitis with polyposis: evaluation with the novel Perioperative Sinus Endoscopy (POSE) scoring system. Laryngoscope. 2007 Nov;117(11 Pt 2 Suppl 115):1-28. doi: 10.1097/MLG.0b013e31814842f8. PMID 18075447
- [Background] Huang Z, Hwang P, Sun Y, Zhou B. Steroid-eluting sinus stents for improving symptoms in chronic rhinosinusitis patients undergoing functional endoscopic sinus surgery. Cochrane Database Syst Rev. 2015 Jun 10;2015(6):CD010436. doi: 10.1002/14651858.CD010436.pub2. PMID 26068957
- [Background] Cote DW, Wright ED. Triamcinolone-impregnated nasal dressing following endoscopic sinus surgery: a randomized, double-blind, placebo-controlled study. Laryngoscope. 2010 Jun;120(6):1269-73. doi: 10.1002/lary.20905. PMID 20513050
- [Background] Smith TL, Singh A, Luong A, Ow RA, Shotts SD, Sautter NB, Han JK, Stambaugh J, Raman A. Randomized controlled trial of a bioabsorbable steroid-releasing implant in the frontal sinus opening. Laryngoscope. 2016 Dec;126(12):2659-2664. doi: 10.1002/lary.26140. Epub 2016 Jul 1. PMID 27363723

RESULTS

PARTICIPANT FLOW:
Groups:
- Bioabsorbable Steroid Releasing Sinus Implant: Patients will undergo bilateral endoscopic sinus surgery which will include bilateral frontal sinusotomy of Draf 2a or 2b type as previously described in the literature. At the conclusion of the procedure, if the patient still meets all inclusion criteria, one frontal sinus will be randomly assigned using the envelop method to receive a bioabsorbable steroid releasing implant and the other frontal sinus will receive a bioabsorbable nasal dressing impregnated with steroid
  Bioabsorbable steroid releasing sinus implant: After completion of indicated frontal sinus surgery, patients will have a bioabsorbable steroid releasing implant placed in the frontal sinus opening, which will remain in place for 14 days.
Period: Overall Study
Arm/Group | Bioabsorbable Steroid Releasing Sinus Implant
Started | 9
Completed | 2
Not Completed | 7
Not completed — Subjects chose not to attend the SOC 12 month follow up visit | 6
Not completed — Clinic was closed due to COVID-19 for 12 month follow up visit | 1

BASELINE CHARACTERISTICS:
Arm/Group | Bioabsorbable Steroid Releasing Sinus Implant
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Whose Propel Sinus Stent Appeared Worse, the Same, or Better Than the Bioabsorbable Nasal Dressing
Description: Grading by a blinded independent sinus expert as to whether the propel sinus stent frontal sinusotomy side is better, worse or the same, in terms of overall appearance after implant removal
Time Frame: 12 months
Population: Two subjects completed the 12 month follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Bioabsorbable Steroid Releasing Sinus Implant & Nasal Dressing Impregnated With Steroid
Number analyzed (Participants) | 2
Participants
  propel sinus stent frontal sinusotomy side is better | 0
  propel sinus stent frontal sinusotomy side is same | 1
  propel sinus stent frontal sinusotomy side is worse | 1

2. Secondary Outcome: Adhesion/Scarring Scale - Left Side
Description: Average adhesion/scarring Likert scale score (range from 0 to 4 with higher numbers indicating worse health) for appearance of the Frontal sinus opening after bioabsorbable steroid releasing implant placement - Left side
Time Frame: 12 months
Population: Data was collected from 3 subjects at 12 months for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Bioabsorbable Steroid Releasing Sinus Implant & Nasal Dressing Impregnated With Steroid
Number analyzed (Participants) | 3
Participants
  adhesion/scarring Likert scale score of 0 | 3
  adhesion/scarring Likert scale score of 1 | 0

3. Secondary Outcome: Adhesion/Scarring Scale - Right Side
Description: Average adhesion/scarring Likert scale score (range from 0 to 4 with higher numbers indicating worse health) for appearance of the Frontal sinus opening after bioabsorbable nasal dressing with added steroid placement
Time Frame: 12 months
Population: Data was collected from 3 subjects at 12 months for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Bioabsorbable Steroid Releasing Sinus Implant & Nasal Dressing Impregnated With Steroid
Number analyzed (Participants) | 3
Participants
  adhesion/scarring Likert scale score of 0 | 2
  adhesion/scarring Likert scale score of 1 | 1

4. Secondary Outcome: Polypoid Edema Scale - Left Side
Description: Average polypoid edema Likert scale score (range from 0 to 4 with higher numbers indicating worse health) for appearance of the Frontal sinus opening after bioabsorbable steroid releasing implant placement
Time Frame: 12 months
Population: Data was collected from 3 subjects at 12 months for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Bioabsorbable Steroid Releasing Sinus Implant & Nasal Dressing Impregnated With Steroid
Number analyzed (Participants) | 3
Participants
  polypoid edema Likert score 0 | 0
  polypoid edema Likert score 1 | 0
  polypoid edema Likert score 2 | 0
  polypoid edema Likert score 3 | 0
  polypoid edema Likert score 4 | 3

5. Secondary Outcome: Polypoid Edema Scale - Right Side
Description: Average polypoid edema Likert scale score (range from 0 to 4 with higher numbers indicating worse health) for appearance of the Frontal sinus opening after bioabsorbable nasal dressing with added steroid placement
Time Frame: 12 months
Population: Data was collected from 3 subjects at 12 months for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Bioabsorbable Steroid Releasing Sinus Implant & Nasal Dressing Impregnated With Steroid
Number analyzed (Participants) | 3
Participants
  polypoid edema Likert score 0 | 1
  polypoid edema Likert score 1 | 0
  polypoid edema Likert score 2 | 0
  polypoid edema Likert score 3 | 0
  polypoid edema Likert score 4 | 2

6. Secondary Outcome: Frontal Sinus Opening Size
Description: Frontal sinus opening greater than or equal to 4 mm for bioabsorbable steroid releasing implant vs. bioabsorbable nasal dressing with added steroid
Time Frame: 12 months
Population: Data was collected from 3 subjects at 12 months for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Bioabsorbable Steroid Releasing Sinus Implant & Nasal Dressing Impregnated With Steroid
Number analyzed (Participants) | 3
Participants
  Left: Yes | 0
  Left: No | 3
  Right: Yes | 1
  Right: No | 2

7. Secondary Outcome: Visualization of Frontal Sinus Roof
Description: Odds ratio of frontal sinus roof visualized for bioabsorbable steroid releasing implant vs. bioabsorbable nasal dressing with added steroid
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Bioabsorbable Steroid Releasing Sinus Implant & Nasal Dressing Impregnated With Steroid
Number analyzed (Participants) | 2
Participants
  Yes | 0
  No | 2

8. Post Hoc Outcome: Number of Participants Whose Propel Sinus Stent Appeared Worse, the Same, or Better Than the Bioabsorbable Nasal Dressing
Description: as for outcome 1
Time Frame: 30 Days
Population: Data was collected from 8 patients at day 30 for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Bioabsorbable Steroid Releasing Sinus Implant & Nasal Dressing Impregnated With Steroid
Number analyzed (Participants) | 8
Participants
  propel sinus stent frontal sinusotomy side is better | 2
  propel sinus stent frontal sinusotomy side is same | 3
  propel sinus stent frontal sinusotomy side is worse | 3

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Bioabsorbable Steroid Releasing Sinus Implant
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-01): https://cdn.clinicaltrials.gov/large-docs/22/NCT03188822/Prot_SAP_000.pdf